CLINICAL TRIAL: NCT06913543
Title: Effect of Open Kinetic Chain Knee Extension Exercises With Neuromuscular Electrical Stimulation in Patients With Post-ACL Reconstruction Surgery
Brief Title: Effect of Open Kinetic CKE Exercises With NES in Patients With Post-ACL Reconstruction Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/806
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental Group - OKC + NMES) (Experimental)
  Interventions: Combination Product: Group 1 (Experimental Group - OKC + NMES)
- Group 2 (Control Group - OKC Only (Active Comparator)
  Interventions: Diagnostic Test: Group 2 (Control Group - OKC Only

INTERVENTIONS:
Combination Product: Group 1 (Experimental Group - OKC + NMES) — OKC Knee Extension Exercises:
  Seated Knee Extensions:
  Resistance bands or machine, 10-15 reps, 2-3 sets.
  Straight Leg Raises:
  With or without ankle weights, 12-15 reps, 2-3 sets.
  Quadriceps Isometric Holds:
  Held for 5-10 seconds, 10 reps, 2-3 sets.
  Neuromuscular Electrical Stimulation (NMES):
  Electrode Placement:
  Over the motor points of the quadriceps.
  Frequency:
  35-50 Hz.
  Pulse Duration:
  200 microseconds.
  Intensity:
  Adjusted for strong yet tolerable contractions.
  On-Off Cycle:
  10 seconds on, 20 seconds off.
  Arms: Group 1 (Experimental Group - OKC + NMES)
Diagnostic Test: Group 2 (Control Group - OKC Only — Open Kinetic Chain Knee Extension Exercises without NMES. Method & Details: The same OKC exercises as the experimental group but without NMES. All exercises are supervised by trained physiotherapists.
  Arms: Group 2 (Control Group - OKC Only

SUMMARY:
"Anterior cruciate ligament (ACL) reconstruction is a commonly performed surgical procedure for restoring knee stability in patients following ACL injuries. Despite surgical success, postoperative rehabilitation remains crucial for improving functional outcomes, addressing quadriceps strength deficits, and reducing recovery time.

DETAILED DESCRIPTION:
This study investigates the combined impact of open kinetic chain (OKC) knee extension exercises and neuromuscular electrical stimulation (NMES) on the functional recovery of post-ACL reconstruction patients. This randomized clinical trial involves 58 patients, divided into two groups: an experimental group receiving OKC knee extension exercises combined with NMES and a control group receiving OKC exercises alone. Functional outcomes, range of motion (ROM), and patient-reported outcomes (PROs) are assessed using validated tools.

ELIGIBILITY:
Inclusion Criteria:

* Both genders aged 18-45 years
* Subjects who have undergone unilateral primary ACL reconstruction surgery
* Subjects who are exactly 4 weeks post-surgery at the start of the study
* Subjects who received a hamstring tendon autograft or patellar tendon graft for ACL reconstruction
* Subjects cleared by a physician to begin open kinetic chain exercises in their rehabilitation program
* Subjects who are generally healthy with no significant comorbidities that could interfere with rehabilitation
* Willingness to provide informed consent and commit to the entire duration of the study

Exclusion Criteria:

* Presence of additional knee injuries (e.g., meniscal tears, collateral ligament injuries) that might affect rehabilitation
* History of prior ACL injury or reconstruction on the same knee
* Patients who underwent reconstruction of other ligaments along with the ACL
* Presence of conditions (e.g., rheumatoid arthritis, osteoarthritis, uncontrolled diabetes) that could influence recovery
* Any significant injury or surgery to the opposite knee within the last six months
* Factors that indicate a high risk of non-compliance with the rehabilitation protocol, such as poor availability, or lack of commitment to follow the exercise regimen
* Conditions affecting neuromuscular control that could interfere with exercise performance or rehabilitation response

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Lysholm Knee Scoring Scale | 12 Months
  Measures knee function with a maximum score of 100.
  Scoring Interpretation:
  95-100 points: Excellent function. 84-94 points: Good function. 65-83 points: Fair function. <65 points: Poor function.
Universal Goniometer | 12 Months
  Measures ROM (Flexion & Extension).
  Interpretation:
  Knee flexion and extension are assessed against standard angles. Higher reliability and validity in measuring knee movement.

CONTACTS AND LOCATIONS:
Locations (1):
- MOVEBETTER 14-A Koh-e-Noor Road, Basement Salt N Pepper, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No